CLINICAL TRIAL: NCT00003961
Title: Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) After T-Lymphocyte Depleted Allogeneic BMT for Myelodysplastic Syndromes
Brief Title: Sargramostim After Bone Marrow Transplantation in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067160, J9852; P30CA006973 (NIH); JHOC-J9852; JHOC-98071505; NCI-G99-1544
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase II trial to study the effectiveness of sargramostim after bone marrow transplantation in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of sargramostim (GM-CSF) on the progression-free 1-year survival of patients with myelodysplastic syndrome who have undergone T-cell-depleted CD34+ augmented allogeneic bone marrow transplantation.

OUTLINE: All patients receive elutriated, CD34+ stem cell augmented donor bone marrow according to another protocol on day 0.

Patients receive sargramostim (GM-CSF) subcutaneously on days 5-60.

Patients are followed on days 120, 180, 360 and periodically thereafter.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically proven myelodysplastic syndrome (MDS) of one of the following types:

  * Refractory anemia with excess blasts (RAEB)
  * RAEB in transformation
  * Chronic myelomonocytic leukemia
  * MDS with multiple chromosomal abnormalities
  * MDS with life threatening cytopenias in at least 2 cell lines

    * Platelet count < 30,000/mm^3 OR
    * Absolute neutrophil count no greater than 1,000/mm^3 OR
    * Anemia requiring transfusion support
  * Leukemia out of MDS (meet any of above requirements, but greater than 30% blasts in marrow)
* No acute leukemia
* Medically eligible for bone marrow transplant according to standard operating procedure of the Sidney Kimmel Cancer Center at Johns Hopkins Blood and Bone Marrow Transplant

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior acute allergic reactions to sargramostim (GM-CSF)
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States